CLINICAL TRIAL: NCT06936696
Title: Project PAIR: Parent-implemented Articulation Intervention With Recast
Acronym: Project PAIR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Meganne Muir, PhD Student and Certified Speech-Language Pathologist, Vanderbilt University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 240777
Record Dates: First submitted 2025-04-13; First posted 2025-04-20 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Hearing Impaired Children
Keywords: deaf and hard of hearing; articulation; speech sound production; parent training; children
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Intervention Model Description: Single case multiple baseline across participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Articulation Therapy (Experimental): Participants engage in two conditions: (1) Parent-implemented Broad Target Speech Recast (BTSR), (2) Parent-implemented BTSR combined with clinician-implemented speech therapy
  This is a nonconcurrent multiple probe single-case experimental design with staggered introduction of conditions across participants. All participants receive both interventions, but the interventions are introduced in separate phases and evaluated independently and in combination.
  This is not a crossover or parallel group design. Rather than having separate arms or randomization, each participant serves as their own control over time, allowing for individualized evaluation of intervention effects.
  Interventions: Behavioral: Broad Target Speech Recast; Behavioral: Traditional Speech Therapy

INTERVENTIONS:
Behavioral: Broad Target Speech Recast — Broad Target Speech Recasts (BTSR) is a speech intervention technique in which an adult immediately recasts a child's incorrect articulation by providing a corrected version of the word in a naturalistic, meaningful context. Unlike traditional articulation therapy, which focuses on isolated sound drills, BTSR integrates correction seamlessly into conversation without requiring the child to repeat or imitate the model.
  This approach is rooted in principles of implicit learning, where repeated exposure to accurate speech models facilitates phonological development over time. BTSR differs from traditional minimal pair or phonetic placement techniques in that it does not involve explicit instruction or direct prompts for self-correction. Instead, it provides high-frequency, naturalistic exposure to correct phoneme production within functional language use.
  Other Names: BTSR
Behavioral: Traditional Speech Therapy — Traditional Speech Therapy is clinician-led and includes structured, drill-based approaches. Techniques such as placement cues, direct feedback, and reinforcement are used to help children achieve correct articulation. The structured nature of this approach is often more effective in remediating persistent speech errors than parent-implemented strategies alone.
  This study examines whether the combination of parent-implemented BTSR and clinician-led traditional articulation therapy leads to improved speech sound production and long-term maintenance of correct articulation in elementary-aged DHH children.

SUMMARY:
Using a single-case multiple baseline across participants design, this study aims to explore the effectiveness of parent-implemented Broad Treatment Speech Recast supplemented with traditional clinician-led articulation therapy on speech production in elementary-aged deaf and hard of hearing children.

To address these objectives, the following research questions will be investigated:

1. Does drill-based articulation therapy, administered by a speech-language pathologist, improve speech sound production in DHH children when parent-implemented BTSR is concurrently utilized at home?
2. Does the combination of parent-implemented BTSR and clinician-led traditional articulation therapy result in generalization of speech sound accuracy at the conversation level?

ELIGIBILITY:
Inclusion Criteria:

* Age 4;0-9;11
* Permanent, prelingual sensorineural hearing loss
* Uses spoken English as their primary home language (≥ 51% of the time)
* Standard score ≥70 on the Leiter
* Standard score ≥70 on the OWLS-II Listening Comprehension
* At least two speech sound errors appropriate to target based on speech norms and general stimulability

Exclusion Criteria:

* Motor speech disorder (e.g., childhood apraxia of speech)
* Oral structural functional disorder (e.g., cleft palate)
* Diagnosis of autism spectrum disorder
* Diagnosis of ADHD
* Uncorrected vision impairment (i.e., identified vision loss without the use of corrective lenses)

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2025-06-10 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Target phoneme production accuracy | From baseline until end of treatment (when intervention criteria have been reached or 6 weeks of no progress / regression)
  The percent of accurate phoneme productions per target, which is derived by dividing the number of correct productions by the total possible points for each target and then multiplying by 100. Accurate phoneme production is defined by a speech-language pathologist's judgment of perceptual accuracy through the lens of broad transcription.

SECONDARY OUTCOMES:
Goldman Fristoe Test of Articulation - Third Edition (GFTA-3) | Collected during eligibility (before the intervention) and at the end of the intervention (when intervention criteria have been reached or 6 weeks of no progress / regression)
  The Goldman-Fristoe Test of Articulation, Third Edition (GFTA-3) is a standardized assessment used to evaluate speech sound production in children, adolescents, and young adults (ages 2;0-21;11). It measures articulation skills by assessing a child's ability to produce consonant sounds in different word positions (initial, medial, final) and in connected speech. The test provides standard scores, percentile ranks, and age-equivalent scores.
  Scores are standardized with a mean of 100 and a standard deviation of 15. Standard scores range from 40 to 160, with higher scores indicating better articulation abilities.
Generalization to Conversation | From enrollment to the end of treatment (when child meets criteria or exhibits no progress/regression for three consecutive sessions).
  Connected speech samples will involve a ten-minute conversation or play-based dialog initiated by the examiner or parent to elicit natural speech from the child. Various techniques may be employed to encourage a sample abundant in expressive language, including the use of open-ended questions and engagement in child-led pretend play. This task will occur at three time-points throughout the study (baseline, BTSR phase, after intervention criteria has been reached) to measure generalization, and it should be administered after the listening check and before the probe. This task will be captured on video for later analysis. Accuracy of phoneme targets will be calculated using percent of consonants correct.

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States